CLINICAL TRIAL: NCT07161947
Title: Shanghai Clinical Cohort-Hyperglycemia in Pregnancy (Reserved)
Brief Title: Shanghai Clinical Cohort of Hyperglycemia in Pregnancy
Acronym: SHINE
Status: Recruiting | Type: Observational
Sponsor: Shanghai General Hospital, China (Other)
Collaborators: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Shanghai First Maternity and Infant Hospital (Other); RenJi Hospital (Other)
Responsible Party: Principal Investigator, Yufan Wang, Chief Physician, Professor, Shanghai General Hospital, China
Other Study IDs: SHDC2025CCS041
Record Dates: First submitted 2025-08-26; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Hyperglycemia in Pregnant Diabetic Patients; Gestatiaonl Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Serum/Plasma, Adipose Tissue, Placenta

SUMMARY:
Establish a high-quality clinical cohort of hyperglycemia in pregnancy. Develop subtype-specific, end-to-end standards for diagnosis, treatment, and follow-up across the preconception, pregnancy, and postpartum phases. These standards will lay a solid foundation for efficient, high-quality clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals who provide written informed consent
* At enrollment, meet one of the following:

  1. Gestational diabetes mellitus (GDM) diagnosed by a 75-g oral glucose tolerance test (OGTT) using Chinese Diabetes Society (CDS) 2024 thresholds (any one of: fasting plasma glucose ≥5.1 mmol/L, 1-h ≥10.0 mmol/L, or 2-h ≥8.5 mmol/L); or 2. Pre-gestational diabetes (type 1 or type 2) documented prior to pregnancy or meeting diabetes criteria at the first prenatal visit (e.g., fasting ≥7.0 mmol/L, 2-h OGTT ≥11.1 mmol/L, or HbA1c ≥6.5%); or 3. At high risk for GDM, defined a priori as ≥1 of the following: prior GDM; prior macrosomic infant (≥4,000 g); pre-pregnancy BMI ≥24 kg/m²; age ≥45 years; high-density lipoprotein cholesterol <1 mmol/L, and/or triglyceride levels >2.8 mmol/L; first-degree family history of diabetes; polycystic ovary syndrome (PCOS); history of coronary heart disease; chronic hypertension and repeated positive fasting urinary glucose in early pregnancy
* Age ≥18 years at the time of consent
* Willing and able to attend postpartum assessments (OGTT at 6 weeks, 12 months, and annually thereafter), with planned follow-up ≥3 years

Exclusion Criteria:

* Current or history of illicit drug use or substance abuse
* Presence of an active infectious disease, including but not limited to: viral hepatitis, sexually transmitted infections or tuberculosis
* Any other condition which, in the judgment of the investigator, would make the subject unsuitable for enrollment in the study

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients who receive routine prenatal care, deliver, and undergo postpartum endocrinology follow-up at any of the following four hospitals: Shanghai General Hospital; Shanghai First Maternity and Infant Hospital; Renji Hospital, Shanghai Jiao Tong University School of Medicine; and Shanghai Sixth People's Hospital Affiliated to Shanghai JiaoTong University.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite Adverse Maternal and Neonatal Outcomes Among Pregnant Individuals With Hyperglycemia in Pregnancy | From delivery (Day 0) through the initial birth hospitalization, assessed up to 14 days postpartum.
  Unit of Measure: Percentage of pregnancies with ≥ 1 event (%) Description: The composite will be coded as Yes/No. An event is counted if any of the following occurs: preeclampsia, cesarean delivery, premature rupture of membranes, placental abruption, preterm birth, congenital malformations, macrosomia, large for gestational age, small for gestational age, neonatal hypoglycemia, neonatal hyperbilirubinemia, neonatal respiratory distress syndrome, neonatal intensive care unit admission, obstetric trauma or still birth. Data abstracted from electronic medical records.
Postpartum Glucose Metabolism Outcomes Among Pregnant Individuals With Hyperglycemia in Pregnancy (OGTT) | From 6 weeks postpartum through long-term follow-up, with assessments at 6 weeks and every 12 months thereafter, for ≥3 years and up to 10 years postpartum.
  Unit of Measure: Percentage of patients with abnormal glucose metabolism based on OGTT (%) Description: This measure will assess the incidence of abnormal glucose metabolism using an oral glucose tolerance test (OGTT). Abnormal glucose metabolism will be defined as: fasting glucose ≥6.1 mmol/L or 2-hour glucose ≥7.8 mmol/L.
  Data will be collected from blood tests and medical records.

SECONDARY OUTCOMES:
Postpartum Glucose Metabolism Outcomes Among Pregnant Individuals With Hyperglycemia in Pregnancy (HbA1c) | From 6 weeks postpartum through long-term follow-up, with assessments at 6 weeks and every 12 months thereafter, for ≥3 years and up to 10 years postpartum.
  Unit of Measure: Percentage of patients with abnormal Hemoglobin A1c (HbA1c, %) Description: This measure will assess the incidence of abnormal glucose metabolism based on HbA1c testing. Abnormal glucose metabolism will be defined as an HbA1c ≥6.5%.
  Data will be collected from blood tests and medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, China, Shanghai, Shanghai Municipality, China